CLINICAL TRIAL: NCT01392599
Title: Surgical Treatment of Complex Regional Pain Syndrome Type II (CRPS II) by Regional Subcutaneous Venous Sympathectomy
Brief Title: Surgical Treatment Of Complex Regional Pain Syndrome Type II (CRPS II)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Wolfgang Happak, Prof. MD, Division of Plastic and Reconstructive Surgery, Surgical Clinic, Medical University of Vienna, Austria
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 026/2009
Record Dates: First submitted 2011-06-30; First posted 2011-07-12 (Estimated); Last update posted 2011-07-12 (Estimated); Status verified 2011-06

CONDITIONS: CRPS Type II
Keywords: CRPS Type II; Pain; Surgery; Regional Subcutaneous Venous Sympathectomy(RSVS); Sudeck; Reflex sympathetic dystrophy (RSD); Causalgia; Algodystrophy
MeSH Terms: conditions — Causalgia; Pain; Reflex Sympathetic Dystrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Surgery (Experimental): Patients with CRPS Type II
  Interventions: Procedure: SUBCUTANEOUS VENOUS SYMPATHECTOMY (RSVS)

INTERVENTIONS:
Procedure: SUBCUTANEOUS VENOUS SYMPATHECTOMY (RSVS) — After incision of the skin a subcutaneous area of approximately 16 cm² (2.5 square inches) will be en block removed between dermis and muscle fascia. All prior detected and marked veins in the operating field will be ligated or coagulated precisely.The tissue defect generated by this operation will be closed by a full thickness or a meshed skin graft which arises during the preparation.

SUMMARY:
The purpose of this study is to investigated and evaluated the effectiveness of a new surgical technique for the treatment of severe chronic pain stages (Complex Regional Pain Syndrome Type II).

DETAILED DESCRIPTION:
For 140 years the treatment of Complex Regional Pain Syndromes Type II (CRPS II) has been an unsolved problem. Recent findings in animal models assume that CRPS Type II is maintained by a coupling of newly sprouted sympathetic and sensible fibres. Therapeutic approaches have included conventional pain medication, physical therapy, sympathetic blocks, transcutaneous or spinal cord stimulation, injections or infusion therapies and sympathectomy. Alone or in combination these therapies often yielded unfavorable results. The majority of physicians dealing with CRPS patients are convinced that a surgical treatment of the affected extremity only exacerbates the symptoms, especially its hallmark excruciating pain.

Patients with a CRPS Type II at the upper or the lower limb will be included in the study after ineffective pain therapy for more than 6 months. The most proximal region of pain associated with CRPS can be localized and 2% Lidocain will be injected into that area. If the sympathetic, deep, burning pain can be blocked repeatedly with these injections, the subcutaneous veins in the previously determined area will be surgically removed. This operation should lead to the permanent resolution of symptoms.

A visual analogue scale (VAS), the Nottingham Health Profile (NHP), thermography and physical examinations will be used to evaluate the outcome of the operation.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from CRPS Type II after after ineffective pain therapy for more than 6 months.

Exclusion Criteria:

* Ineffective testinfiltration with an local anesthetic Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-01; Primary Completion 2013-01 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Enhancement in the quality of life (measured by the NHP) due to a permanent reduction of pain (measured by the NHP and a VAS) of patients suffering from CRPS Type II. | Outcome measures will be evaluated at baseline and 6 weeks after the operation
  An appraisal of results will be made after the operation by using physical examionations and the standardized questionnaires (NHP,VAS). The health status and especially the pain level have to be constant for at least 3 month before being considered as an result.

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Happak, Prof. MD, Principal Investigator — Division of Plastic and Reconstructive Surgery, Department of Surgery, Medical University of Vienna, Austria
Locations (1):
- Division of Plastic and Reconstructive Surgery, Department of Surgery, Medical University of Vienna, Vienna, Vienna, Austria

REFERENCES:
- [Background] Bruehl S, Harden RN, Galer BS, Saltz S, Bertram M, Backonja M, Gayles R, Rudin N, Bhugra MK, Stanton-Hicks M. External validation of IASP diagnostic criteria for Complex Regional Pain Syndrome and proposed research diagnostic criteria. International Association for the Study of Pain. Pain. 1999 May;81(1-2):147-54. doi: 10.1016/s0304-3959(99)00011-1. PMID 10353502
- [Background] Albrecht PJ, Hines S, Eisenberg E, Pud D, Finlay DR, Connolly KM, Pare M, Davar G, Rice FL. Pathologic alterations of cutaneous innervation and vasculature in affected limbs from patients with complex regional pain syndrome. Pain. 2006 Feb;120(3):244-266. doi: 10.1016/j.pain.2005.10.035. Epub 2006 Jan 19. PMID 16427199
- [Background] Oaklander AL, Rissmiller JG, Gelman LB, Zheng L, Chang Y, Gott R. Evidence of focal small-fiber axonal degeneration in complex regional pain syndrome-I (reflex sympathetic dystrophy). Pain. 2006 Feb;120(3):235-243. doi: 10.1016/j.pain.2005.09.036. Epub 2006 Jan 19. PMID 16427737
- [Background] Arnold JM, Teasell RW, MacLeod AP, Brown JE, Carruthers SG. Increased venous alpha-adrenoceptor responsiveness in patients with reflex sympathetic dystrophy. Ann Intern Med. 1993 Apr 15;118(8):619-21. doi: 10.7326/0003-4819-118-8-199304150-00008. No abstract available. PMID 8383935
- [Background] Baron R, Schattschneider J, Binder A, Siebrecht D, Wasner G. Relation between sympathetic vasoconstrictor activity and pain and hyperalgesia in complex regional pain syndromes: a case-control study. Lancet. 2002 May 11;359(9318):1655-60. doi: 10.1016/S0140-6736(02)08589-6. PMID 12020526
- [Background] Drummond PD, Finch PM, Smythe GA. Reflex sympathetic dystrophy: the significance of differing plasma catecholamine concentrations in affected and unaffected limbs. Brain. 1991 Oct;114 ( Pt 5):2025-36. doi: 10.1093/brain/114.5.2025. PMID 1933231